CLINICAL TRIAL: NCT04637919
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Clinical Trial to Investigate the Safety and Immunogenicity of High-dose IN-B001 After Administration in Healthy Subjects
Brief Title: Safety and Immunogenicity of High-dose IN-B001 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IN_HFM_102
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Hand, Foot and Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IN-B001 EV71 A dose (Experimental): Inactivated EV71 vaccine(A dose) or placebo in 10 healthy adults (three doses, 28 days interval)
  Interventions: Biological: IN-B001 EV71 A dose; Biological: Placebo
- IN-B001 CVA16 B dose (Experimental): Inactivated CVA16 vaccine(B dose) or placebo in 10 healthy adults (three doses, 28 days interval)
  Interventions: Biological: IN-B001 CVA16 B dose; Biological: Placebo
- IN-B001 Bivalent C dose (Experimental): Inactivated EV71/CVA16 vaccine(C dose) or placebo in 10 healthy adults (three doses, 28 days interval)
  Interventions: Biological: IN-B001 Bivalent C dose; Biological: Placebo

INTERVENTIONS:
Biological: IN-B001 EV71 A dose — Inactivated vaccine against EV71, three doses, 28 days interval
  Arms: IN-B001 EV71 A dose
Biological: IN-B001 CVA16 B dose — Inactivated vaccine against CVA16, three doses, 28 days interval
  Arms: IN-B001 CVA16 B dose
Biological: IN-B001 Bivalent C dose — Inactivated vaccine against EV71/CVA16, three doses, 28 days interval
  Arms: IN-B001 Bivalent C dose
Biological: Placebo — Placebo, three doses, 28 days interval

SUMMARY:
This study aims to evaluate the safety and immunogenicity of high-dose IN-B001 after administration in healthy subjects

DETAILED DESCRIPTION:
Enterovirus 71(EV71) and coxsackievirus A16(CVA16) are major causes of Hand-foot-and-mouth disease (HFMD) occurring in pediatric population. Although EV71 vaccine has been licensed in China, vaccine for CVA16-associated HFMD is currently not available anywhere. The purpose of this phase I study is to evaluate the safety and immunogenicity of EV71/CVA16 bivalent vaccine in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged ≥19 to <50 years at the time of screening tests
* Body mass index(BMI) of ≥18.0 kg/m2 to ≤27.0 kg/m2, with body weight of ≥55.0 kg to ≤90.0 kg for men and ≥50.0 kg to ≤90.0 kg for women at the time of screening tests
* Determined by the investigator to be eligible for study participation based on the results of screening tests
* Intact deltoid muscle that allows administration of the investigational product
* Consent to use medically acceptable contraception throughout the study
* Negative finding from a pregnancy test (urine hCG) at the time of the screening for women of childbearing potential
* Voluntary decision and provision of written consent on participation in this study

Exclusion Criteria:

* History of a hand-foot-mouth disease or history of a disease related with enterovirus(EV) infection within 3 months prior to the 1st IP administration
* Medical history of an anaphylactic or similar acute reaction to IN-B001 or similar vaccine
* Febrile disease or infectious disease within 2 weeks prior to the 1st IP administration
* Whole blood donation within 2 months or apheresis within 1 month prior to the 1st IP administration
* Vaccination with other prevention vaccine within 2 months prior to the 1st IP administration
* Use of an immunomodulator or immunosuppressant within 3 months prior to the 1st IP administration
* History of a Guillain Barre syndrome
* Excessive caffeine intake or continuous alcohol consumption or incapable of abstention from alcohol during the study
* Participation in other clinical trial within 6 months prior to the 1st IP administration
* Pregnant or breastfeeding women
* Clinically significant hepatic, renal, neurological, respiratory, endocrine, hematology and oncology, cardiovascular, urological or psychiatric disease or such history
* Positive serological finding (type B hepatitis test, type C hepatitis test, human immunodeficiency virus(HIV) test)
* History of drug abuse or positive finding from a urine screening test for an abusive drug
* Use or of any prescription medication or oriental medicine within 2 weeks or any over-the-counter(OTC) medication, health functional food or vitamin within 1 week prior to the 1st IP administration or expected use of such products
* Administration of a blood product or blood-derived agent within 3 months prior to the 1st IP administration
* Determined by the investigator to be ineligible for study participation due to other reason including clinical laboratory findings

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events of IN-B001 (Safety of IN-B001) | Week 0 to Week 32
  Frequency and severity of adverse events up to 32 weeks post first dose

SECONDARY OUTCOMES:
Immunogenicity of IN-B001: Anti-EV71 IgG titer | Week 0 to Week 32
  Serum EV71-specific IgG titers
Immunogenicity of IN-B001 : Anti-CVA16 IgG titer | Week 0 to Week 32
  Serum CVA16-specific IgG titers
Immunogenicity of IN-B001 : Geometric mean titer (GMT) of EV71 neutralizing antibody titers | Week 0 to Week 32
  Geometric mean titers based on neutralizing antibody titers. Measurement of fold-increase over baseline of neutralizing titers against EV71
Immunogenicity of IN-B001 : GMT of CVA16 neutralizing antibody titers | Week 0 to Week 32
  Geometric mean titers based on neutralizing antibody titers. Measurement of fold-increase over baseline of neutralizing titers against CVA16

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, Ph.D, Principal Investigator — Seoul National University Hospital, Dept. of Clinical Pharmacology
Locations (1):
- Seoul National University Hospital, Clinical Trial Center, Seoul, South Korea